CLINICAL TRIAL: NCT00236951
Title: A Phase III Randomized Controlled Study Comparing Iron Sucrose Intravenously to No Iron Treatment of Anemia in Cancer Patients Undergoing Chemotherapy and Erythropoietin Therapy
Brief Title: Intravenous (IV) Iron vs. No Iron as the Treatment of Anemia in Cancer Patients Undergoing Chemotherapy and Erythropoietin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Marc Tokars, Senior Director of Clinical Operations, Luitpold Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1VEN02023
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: Anemia; Cancer; Chemotherapy
MeSH Terms: conditions — Anemia; Neoplasms

ARMS (4):
- Venofer + erythropoietin (responders) (Active Comparator)
  Interventions: Drug: iron sucrose injection USP
- erythropoietin only (responders) (Active Comparator)
  Interventions: Drug: stable erythropoietin therapy
- Venofer+erythropoietin(non-responders) (Active Comparator)
  Interventions: Drug: iron sucrose injection USP
- erythropoietin only (non-responders) (Active Comparator)
  Interventions: Drug: stable erythropoietin therapy

INTERVENTIONS:
Drug: iron sucrose injection USP
  Arms: Venofer + erythropoietin (responders); Venofer+erythropoietin(non-responders)
Drug: stable erythropoietin therapy
  Arms: erythropoietin only (non-responders); erythropoietin only (responders)

SUMMARY:
To assess the change in hemoglobin levels when iron sucrose was added to a regimen of weekly, fixed doses of erythropoietin in patients who had or had not responded to erythropoietin therapy alone.

DETAILED DESCRIPTION:
This was a two stage, randomized, controlled study of cancer patients undergoing or planning to undergo chemotherapy. After stage one, (where patients were exposed to an erythropoiesis stimulating agent), patients were randomized to receive either IV iron sucrose or no iron supplementation. Patients were then followed to safety and efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Histological Diagnosis of Cancer
* Hgb </= 10
* Ongoing or Planned Chemotherapy
* Body Weight >50kg
* Free of Active Infection
* Karnofsky Status 60% to 100%

Exclusion Criteria:

* Active infection
* Use of Multivitamins with iron within one week of entry
* Myelophthisic bone marrow involvement by tumor except hematologic malignancy
* Concurrent medical condition that would prevent compliance or jeopardize the health of the patient
* Use of any IV iron products within two months of study entry
* Blood Transfusions
* Hypoplastic bone marrow failure state
* Acute Leukemia
* Myeloproliferative syndrome
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2003-02; Primary Completion 2005-10 (Actual); Study Completion 2005-12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 18, 2003 - October 27, 2005 Locations: Hospitals and Medical Clinics (33 total sites)
Pre-assignment Details: Anemia defined as a hemoglobin level < or = to 10.0 g/dL.
Groups:
- Group A: Erythropoietin + Venofer (Responders): Subjects who at any time during Stage 1 (8-week duration) showed a > or = 1 g/dL increase in hemoglobin over baseline. These subjects received 100mcg of weekly Erythropoietin and up to three 500mg doses of Venofer at intervals of 2 to 3 weeks with last dose no later than Week 9 of Stage 2.
- Group B: Erythropoietin Only (Responders): Subjects who at any time during Stage 1 (8-week duration) showed a > or = 1 g/dL increase in hemoglobin over baseline. These subjects received 100mcg of weekly Erythropoietin only.
- Group C: Erythropoietin + Venofer (Non-responders): Subjects whose maximum hemoglobin increase was < 1 g/dL over baseline were designated as Stage 1 (8-week duration) non-responders. These subjects received 100mcg of weekly Erythropoietin and up to three 500mg doses of Venofer at intervals of 2 to 3 weeks with last dose no later than Week 9 of Stage 2.
- Group D: Erythropoietin Only (Non-responders): Subjects whose maximum hemoglobin increase was < 1 g/dL over baseline were designated as Stage 1 (8-week duration) non-responders. These subjects received 100mcg of weekly Erythropoietin only.
Period: Overall Study
Arm/Group | Group A: Erythropoietin + Venofer (Responders) | Group B: Erythropoietin Only (Responders) | Group C: Erythropoietin + Venofer (Non-responders) | Group D: Erythropoietin Only (Non-responders)
Started | 59 | 77 | 40 | 48
Completed | 33 | 46 | 21 | 17
Not Completed | 26 | 31 | 19 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Erythropoietin + Venofer (Responders) | Group B: Erythropoietin Only (Responders) | Group C: Erythropoietin + Venofer (Non-responders) | Group D: Erythropoietin Only (Non-responders) | Total
Number analyzed (Participants) | 59 | 77 | 40 | 48 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 42 | 23 | 25 | 124
  >=65 years | 25 | 35 | 17 | 23 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 49 | 28 | 31 | 147
  Male | 20 | 28 | 12 | 17 | 77

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Maximum Hemoglobin Level During Stage 2 (Week 9 Through Week 21).
Description: The hemoglobin baseline was defined as the average of the last 2 hemoglobin values during stage 1 (through week 8).
Time Frame: During Stage 2 (week 9 through week 21)
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Group A: Erythropoietin + Venofer (Responders) | Group B: Erythropoietin Only (Responders) | Group C: Erythropoietin + Venofer (Non-responders) | Group D: Erythropoietin Only (Non-responders)
Number analyzed (Participants) | 59 | 77 | 40 | 48
g/dL | 2.6 (1.59) | 1.8 (1.39) | 2.5 (1.88) | 1.3 (1.73)

ADVERSE EVENTS:
Time Frame: 2 years and 3 months
Arm/Group | Group A: Erythropoietin + Venofer (Responders) | Group B: Erythropoietin Only (Responders) | Group C: Erythropoietin + Venofer (Non-responders) | Group D: Erythropoietin Only (Non-responders)
Serious Adverse Events (participants affected / at risk) | 13/59 | 14/77 | 11/40 | 11/48
Other Adverse Events (participants affected / at risk) | 50/59 | 48/77 | 32/40 | 35/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Erythropoietin + Venofer (Responders) (N=59) | Group B: Erythropoietin Only (Responders) (N=77) | Group C: Erythropoietin + Venofer (Non-responders) (N=40) | Group D: Erythropoietin Only (Non-responders) (N=48)
Abdominal Pain NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis acute NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity NOS (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia NOS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral neuropathy NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia NOS (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Resection of Rectum (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis NOS (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Erythropoietin + Venofer (Responders) (N=59) | Group B: Erythropoietin Only (Responders) (N=77) | Group C: Erythropoietin + Venofer (Non-responders) (N=40) | Group D: Erythropoietin Only (Non-responders) (N=48)
Abdominal pain NOS (Gastrointestinal disorders) | 5 (5) | 3 (4) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 4 (4) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
Appetite decreased NOS (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (7) | 3 (3) | 2 (2)
Asthenia (General disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 3 (3) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Canidal infection NOS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Chest pain (General disorders) | 4 (5) | 3 (4) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (8) | 7 (7) | 4 (4) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 0 (0) | 4 (6)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Diarrhea NOS (Gastrointestinal disorders) | 8 (8) | 9 (10) | 6 (6) | 6 (9)
Dizziness (Nervous system disorders) | 6 (6) | 3 (4) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (7) | 8 (8) | 1 (1) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (4) | 3 (4) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (9) | 16 (17) | 6 (8) | 11 (12)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 4 (4) | 4 (6) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 1 (1) | 2 (2)
Hypotension NOS (Vascular disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (22) | 16 (21) | 10 (10) | 8 (10)
Oedema NOS (General disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 7 (7) | 6 (6) | 4 (5) | 2 (2)
Pain NOS (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Peripheral neuropathy NOS (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Rash NOS (Skin and subcutaneous tissue disorders) | 3 (4) | 6 (8) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0) | 4 (4)
Upper respiratory infection NOS (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Vomiting NOS (Gastrointestinal disorders) | 12 (14) | 11 (14) | 5 (7) | 6 (6)
Weight decreased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less